CLINICAL TRIAL: NCT00926172
Title: Epidemiology of Cerebral Aneurysms With MRA in China in Middle-aged or Elder Person: a Population-based Survey
Brief Title: Screening Intracranial Aneurysms With Magnetic Resonance Angiography (MRA) in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Cerebral aneurysm study in China, The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University
Other Study IDs: CASC1; SAPH001
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-12

CONDITIONS: Intracranial Aneurysm
Keywords: Magnetic resonance angiography; Intracranial aneurysm; cerebral aneurysm; unruptured aneurysm; Epidemiology; Magnetic Resonance Imaging
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Chinese Cerebral Aneurysms Survey is a continuing prospective study among middle-aged and older individuals (35 - 75 years) that aims to determine the prevalence of cerebral intracranial aneurysms in the general population with MRA at 3.0 Tesla (T).

DETAILED DESCRIPTION:
Cerebral intracranial aneurysms are common. In angiographic and autopsy studies, estimates for prevalence vary between 0.2 and 9.9 percent. The methods used to detect the aneurysms markedly influenced the proportion of aneurysms. Retrospective autopsy studies probably give an underestimation and prospective angiography studies an overestimation of the actual prevalence. Accurate data on the prevalence of intracranial aneurysms are essential in evaluating the results of screening programs for aneurysms in general population.

During the past decade, MRA, as a preferred accuracy modality for noninvasive intracranial vascular imaging at most centers, is playing an increasing role in the evaluation of patients suspected of having intracranial aneurysms. In recurrent study, we have tested that MRA at 3T has excellent sensitivity, accuracy, and correlation with DSA and is comparable to catheter cerebral angiography for the evaluation of patients with intracranial aneurysms (Stroke, in press). Therefore, we examined trends in intracranial aneurysm prevalence with the use of MRA at 3.0T to determine the true prevalence of cerebral intracranial aneurysms in the general middle-aged or elder population.

ELIGIBILITY:
Inclusion Criteria:

* Native inhabitants lived in a defined area sites in China
* Aged 35-75 years

Exclusion Criteria:

* Less than 35 years old or more than 75 years old
* Incompetent patient who cannot give consent for routine MR Angiography and his/her surrogate decision maker is not available
* Any patients with a contraindication to having a standard MRI examination, such as phase maker, orbital metallic foreign body, etc.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators recruited 4500-5000 native inhabitants aged 35-75 years lived in China according to China census-tract data from the year 2005. The gender was accordance with China census-tract data, and the population aged 35-75 years has a higher incident of intracranial aneurysm in the literature. Assuming an 8 percent prevalence of intracranial aneurysm in the general population and using a two-sided alpha value of 0.05, the investigators estimated that 4500-5000 native inhabitants would need to be enrolled for the study.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Cerebral intracranial aneurysms identified by 3-D TOF-MRA at 3T | 18 months after the study

SECONDARY OUTCOMES:
Suspected cerebral aneurysms detected by MRA underwent digital subtraction angiography (DSA) examination | 32-36 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hua Li, MD, PhD, Study Chair — The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University; Yong-Dong Li, MD, PhD, Principal Investigator — The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University
Locations (1):
- The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li MH, Cheng YS, Li YD, Fang C, Chen SW, Wang W, Hu DJ, Xu HW. Large-cohort comparison between three-dimensional time-of-flight magnetic resonance and rotational digital subtraction angiographies in intracranial aneurysm detection. Stroke. 2009 Sep;40(9):3127-9. doi: 10.1161/STROKEAHA.109.553800. Epub 2009 Jun 25. PMID 19556531